CLINICAL TRIAL: NCT02662582
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled, Two Period, Crossover Study to Assess the Effect of CK-2127107 on Physical Function in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Assess the Effect of CK-2127107 on Physical Function in Subjects With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Cytokinetics (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3318-CL-3002
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; CK-2127107; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — reldesemtiv

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CK-2127107 1000 mg, then placebo (Experimental): Participants received CK-2127107 500 milligram (mg), orally, twice daily for 2 weeks in treatment period 1 followed by matching placebo orally, twice daily for 2 weeks in treatment period 2. A washout period of 2 weeks was maintained between the two treatment periods.
  Interventions: Drug: Reldesemtiv; Drug: Placebo
- Placebo, then CK-212710 1000 mg (Experimental): Participants received matching placebo orally, twice daily for 2 weeks in treatment period 1 followed by CK-2127107 500 mg in treatment period 2. A washout period of 2 weeks was maintained between the two treatment periods.
  Interventions: Drug: Reldesemtiv; Drug: Placebo

INTERVENTIONS:
Drug: Reldesemtiv — Oral tablet
  Other Names: CK-2127107
Drug: Placebo — Oral tablet

SUMMARY:
The purpose of this study was to assess the effect of CK-2127107 relative to placebo on cycle ergometer exercise tolerance, assessed as change from period baseline in constant work rate (CWR) endurance time, utilizing a breath-by-breath metabolic measurement system with integrated electrocardiogram (ECG). The time to intolerance was assessed by a stopwatch and verified from electronic recordings of the cycle ergometer.

This study assessed cardiopulmonary and neuromuscular effects of CK-2127107 relative to placebo; the effect of CK-2127107 on resting spirometry relative to placebo; the safety and tolerability of CK-2127107 as well as the pharmacokinetics of CK-2127107.

DETAILED DESCRIPTION:
Enrolled participants were randomly assigned to 1 of 2 treatment sequences and received both CK-2127107 and matching placebo over 2 treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) of 18-35 kg/m2 inclusive.
* Subject must have all of the following:

  * Clinical diagnosis of moderate to severe COPD, with a postbronchodilator FEV1/FVC ratio < 70% and 30% ≤ FEV1 < 65% predicted at screening. The predicted values for normal spirometry will be those recommended by the American Thoracic Society (ATS) / European Respiratory Society (ERS) [Miller et al, 2005].
  * General stable health with no change in medication (including non-COPD agents and dietary aids/food supplements) within 2 weeks prior to screening, no systemic corticosteroid administration (topical or inhaled corticosteroids are allowed) within 6 weeks prior to screening, no exacerbations or hospitalization within 6 weeks prior to screening.
  * Current or ex-smokers with a smoking history of at least 10 pack years.
  * Grade of 2 or 3 on the Modified Medical Research Council (mMRC) Dyspnea Scale at screening:

    1. Grade 2: walks slower than people of the same age on the level because of breathlessness or has to stop for breath when walking at own pace on the level.
    2. Grade 3: stops for breath after walking about 100 meters or after a few minutes on the level.
* Subject is able to complete technically acceptable respiratory muscle strength tests, spirometry, physical performance test and exercise tests.
* Female subject must either:

  * Be of non-child bearing potential: Postmenopausal (defined as at least 1 year without any menses) prior to screening, or documented surgically sterile.
  * Or, if of childbearing potential: Agree not to try to become pregnant during the study and for 28 days after the last dose, and have a negative serum pregnancy test at screening, and, if heterosexually active, agree to consistently use 2 forms of highly-effective birth control (at least 1 of which must be a barrier method) starting at screening, throughout the study, and for 28 days after the last dose.
* Female subject must agree not to breastfeed starting at screening and throughout the study and for 28 days after the last dose.
* Female subject must not donate ova starting at screening, throughout the study and for 28 days after the last dose.
* Male subject and their female spouse/partners who are of childbearing potential must be using highly effective form of contraception consisting of 2 forms of birth control (at least 1 of which must be a barrier method) starting at screening, and continuing throughout the study and for 90 days after the last dose.
* Male subject must not donate sperm starting at screening, throughout the study and for 90 days after the last dose.
* Subject agrees not to participate in another interventional study from screening through the follow-up visit (FUV) of the study.

Exclusion Criteria:

* Subject has previously enrolled in a clinical study of CK-2127107.
* Subject has any clinically significant abnormality following the investigator's review of the physical examination, ECG and protocol-defined clinical laboratory tests at screening. A significant abnormality is defined as an abnormality which, in the opinion of the investigator, may (i) put the subject at risk because of participation in the study, (ii) influence the results of the study or (iii) cause concern regarding the subject's ability to participate in the study.
* Subject has any of the liver function tests (LFTs; i.e., aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase [ALP], γ-glutamyl transferase [GGT] and/or total bilirubin [TBL]) above 1.5 times the upper limit of normal (ULN) at screening. These assessments may be repeated once at the investigator's discretion (within the screening window).
* Subject has an estimated glomerular filtration rate (eGFR) less than 30 mL/min/1.73 m2 by the Cockcroft-Gault equation at screening.
* Subject has a serious cardiovascular disease, including a current New York Heart Association (NYHA) class III or IV congestive heart failure or clinically significant valvular disease, history of cardiac arrest, uncontrolled angina or arrhythmia, untreated serious conduction disorder (e.g., third-degree heart block), or acute myocardial ischemic condition suspected on the ECG at screening (e.g., ST-segment elevation, ST-segment depressions > 2 mm).
* Subject has had a myocardial infarction or other acute coronary syndrome, major heart surgery (i.e., valve replacement or bypass surgery), stroke, deep vein thrombosis or pulmonary embolus in the 6 months prior to screening.
* Subject has known active tuberculosis.
* Subject has undergone thoracotomy with pulmonary resection (except for sub-lobar resection).
* Subject has resting pulse < 40 bpm or > 100 bpm; resting systolic blood pressure > 160 mm Hg or < 90 mm Hg; resting diastolic blood pressure > 100 mm Hg at screening. These assessments may be repeated once at the investigator's discretion (within the screening window).
* Subject desaturates to SpO2 < 85% for at least 1 minute on screening IET.
* Subject has a limitation of exercise performance as a result of factors other than fatigue or exertional dyspnea/shortness of breath (considered to be due to COPD), such as arthritis in the leg, angina pectoris, heart failure, claudication or morbid obesity.
* Subject has a CWR cycle ergometry endurance time less than 4 or greater than 8 minutes after WR adjustment procedures.
* Subject has used the following drugs within 14 days prior to day -1:

  * Strong cytochrome P450 (CYP)3A4 inhibitor (e.g., itraconazole, clarithromycin).
  * Strong CYP3A4 inducer (e.g., barbiturates, rifampin).
* Subject has hemoglobin (Hb) concentration below 10.0 g/dL at screening.
* Subject has a cancer requiring treatment currently or in the past 3 years (except primary nonmelanoma skin cancer, carcinoma in situ or cancers that have an excellent prognosis such as early stage breast or prostate cancer).
* Subject giving a history of asthma, allergic rhinitis or atopy shall be evaluated by the investigator to determine whether the subject's predominant diagnosis is COPD rather than asthma.
* Subject has neurological conditions or neuromuscular diseases that are causing impaired muscle function or mobility.
* Subject has a current diagnosis of schizophrenia, other psychotic disorders or bipolar disorder.
* Subject in the active phase of pulmonary rehabilitation or had completed pulmonary rehabilitation or exercise training within the 13 weeks prior to screening.
* Subject has severe and/or uncontrolled medical conditions that could interfere with the study (e.g., severe neurological deficit after stroke, developed diabetic peripheral neuropathy, respiratory diseases requiring daytime supplemental oxygen, infection, gastrointestinal disorder, uncontrolled pain or any other non-stable illness) as judged by the medical investigator.
* Subject has a known history of positive test for hepatitis B surface antigen (HBsAg) or hepatitis C antibody or history of a positive test for human immunodeficiency virus (HIV) infection.
* Subject has a history of alcoholism or drug/chemical substance abuse within 2 years prior to screening.
* Subject has used any medications known to affect physical function or muscle mass including androgen supplements, anti-androgens (such as luteinizing hormone-releasing hormone [LHRH] agonists), anti-estrogen (tamoxifen, etc.), recombinant human growth hormone (rhGH), insulin, oral beta adrenergic agonists, megestrol acetate, dronabinol, metformin or other drugs which, in the opinion of the investigator, might influence physical function or muscle mass within 6 weeks prior to screening.
* Subject has participated in any interventional clinical study or has been treated with any investigational drugs within 28 days or 5 half-lives whichever is longer, prior to the initiation of screening.
* Subject has any other condition that in the opinion of the investigator precludes the subject's participation in the trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (2):
- United States (2):
  - Site US10001, Torrance, California
  - Site US10003, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=379

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with a clinical diagnosis of moderate to severe chronic obstructive pulmonary disease (COPD) between 40 to 75 years of age inclusive and met all of the inclusion and none of the exclusion criteria were enrolled in this study.
Groups:
- CK-2127107 1000 mg, Then Placebo: Participants received CK-2127107 500 mg, orally, twice daily for 2 weeks in treatment period 1 followed by matching placebo orally, twice daily for 2 weeks in treatment period 2. A washout period of 2 weeks was maintained between the two treatment periods.
- Placebo, Then CK-212710 1000 mg: Participants received matching placebo orally, twice daily for 2 weeks in treatment period 1 followed by CK-2127107 500 mg orally, twice daily for 2 weeks in treatment period 2. A washout period of 2 weeks was maintained between the two treatment periods.
Period: Treatment Period 1 (14 Days)
Arm/Group | CK-2127107 1000 mg, Then Placebo | Placebo, Then CK-212710 1000 mg
Started | 23 | 23
Completed | 18 | 19
Not Completed | 5 | 4
Not completed — Adverse Event | 3 | 2
Not completed — Miscellaneous | 0 | 1
Not completed — Protocol Deviation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Period: Washout Period (14 Days)
Arm/Group | CK-2127107 1000 mg, Then Placebo | Placebo, Then CK-212710 1000 mg
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0
Period: Treatment Period 2 (14 Days)
Arm/Group | CK-2127107 1000 mg, Then Placebo | Placebo, Then CK-212710 1000 mg
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAF) consisted of all randomized participants who took ≥ 1 dose of study medication.
Groups:
- CK-2127107 1000mg, Then Placebo: Participants received CK-2127107 500 mg, orally, twice daily for 2 weeks in treatment period 1 followed by matching placebo orally, twice daily for 2 weeks in treatment period 2. A washout period of 2 weeks will be maintained between the two treatment periods.
- Placebo, Then CK-2127107 1000mg: Participants received matching placebo orally, twice daily for 2 weeks in treatment period 1 followed by CK-2127107 500 mg, orally, twice daily for 2 weeks in treatment period 2. A washout period of 2 weeks will be maintained between the two treatment periods.
- Total: Total of all reporting groups
Arm/Group | CK-2127107 1000mg, Then Placebo | Placebo, Then CK-2127107 1000mg | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (7.9) | 63.1 (8.3) | 63 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 23 | 22 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 18 | 14 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Constant work rate (CWR) Endurance Time [Mean (Standard Deviation); unit: Seconds] — The CWR defines how long it takes until the participant reaches symptom limitations while simultaneously being monitored and is called "CWR time to intolerance," which determines the "CWR endurance time".
  Seconds | 334.5 (80.0) | 346.4 (89.1) | 340.4 (84.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Period Baseline at Week 2 in Constant Work Rate (CWR) Endurance Time Relative to Placebo
Description: The CWR defines how long it takes until the participant reaches symptom limitations while simultaneously being monitored and is called "CWR time to intolerance," which determined the "CWR endurance time". Positive change indicates an improvement from baseline (i.e., a favorable outcome).
Time Frame: Baseline and week 2 of each treatment period
Population: The full analysis set (FAS) consisted of all participants who were randomized and received ≥ 1 dose of study drug and had ≥ 1 baseline measurement and 1 post baseline measurement within a period. FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: seconds
Groups:
- Placebo: Participants received matching placebo orally, twice daily for 2 weeks in treatment periods 1 and 2.
- CK-2127107: Participants received CK-2127107 500 mg orally twice daily for 2 weeks in treatment periods 1 and 2.
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
seconds | -1.4 (22.2) | -13.4 (21.2)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; Least square means (LSMeans), LSMean difference of CK-2127107 minus placebo, and 90% confidence intervals are based on a mixed effect model with treatment and period as fixed effects, subject as a random effect, and a compound symmetry covariance structure; Test type: Superiority; p = 0.734, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = -12.0, 90% CI 2-sided [-71.2 to 47.2]

2. Secondary Outcome: Change From Period Baseline at Week 2 in Oxygen Uptake (VO2)
Description: VO2 was defined as volume of O2 extracted from inspired air in a given period of time. VO2 was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Liter per minute (L/min)
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
Liter per minute (L/min)
  Peak | -0.0054 (0.0193) | -0.0273 (0.0182)
  Isotime | -0.0006 (0.0155) | -0.0330 (0.0147)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; Peak: LSMeans, LSMean difference of CK-2127107 minus placebo, and 90% confidence intervals are based on a mixed effect model with treatment and period as fixed effects, subject as a random effect, and a compound symmetry covariance structure; Test type: Superiority; p = 0.438, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean Difference = -0.0219, 90% CI 2-sided [-0.0694 to 0.0256]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; Isotime: LSMeans, LSMean difference of CK-2127107 minus placebo, and 90% confidence intervals are based on a mixed effect model with treatment and period as fixed effects, subject as a random effect, and a compound symmetry covariance structure; Test type: Superiority; p = 0.114, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean Difference = -0.0325, 90% CI 2-sided [-0.0663 to 0.0014]

3. Secondary Outcome: Change From Period Baseline at Week 2 in Ventilation (VE)
Description: VE was defined as volume of gas exhaled from the lungs in 1 minute, also called 'ventilation' or 'minute ventilation. VE was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
L/min
  Peak | -0.17 (1.04) | 0.58 (0.98)
  Isotime | 0.04 (0.84) | 0.34 (0.80)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.612, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.75, 90% CI 2-sided [-1.75 to 3.24]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.789, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.29, 90% CI 2-sided [-1.55 to 2.14]

4. Secondary Outcome: Change From Period Baseline at Week 2 in Ventilatory Equivalent for Carbon Dioxide (VE/VCO2)
Description: VE/VCO2 was a ratio of VE to VCO2. It is a dimensionless quantity. This ratio indicates how many liters of air exhaled were breathed to eliminate 1 liter of CO2. VE/VCO2 was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
ratio
  Peak | 0.05 (0.37) | 0.77 (0.36)
  Isotime | 0.05 (0.37) | 0.97 (0.35)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.225, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.72, 90% CI 2-sided [-0.26 to 1.70]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.064, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.92, 90% CI [0.11 to 1.174]

5. Secondary Outcome: Change From Period Baseline at Week 2 in Inspiratory Capacity (IC) Change From Peak to Rest
Description: IC was defined as the volume of air that can be inspired after a normal expiration; it is the sum of the tidal volume (VT) and the IRV.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
Liters | -0.008 (0.051) | 0.044 (0.048)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; LSMeans, LSMean difference of CK-2127107 minus placebo, and 90% confidence intervals are based on a mixed effect model with treatment and period as fixed effects, subject as a random effect, and a compound symmetry covariance structure; Test type: Superiority; p = 0.447, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.052, 90% CI 2-sided [-0.063 to 0.167]

6. Secondary Outcome: Change From Period Baseline at Week 2 in Perceived Exertion for Dyspnea and Leg Discomfort (BORG CR10)
Description: The Borg Scale (Borg CR10) is a simple 10-item method of rating perceived exertion and collects information on perceived exertion in an individual's rating of exercise intensity. Participants were asked to use this scale to rate the intensity of their breathing and leg discomfort before, during, and after exercise. Scores range from 0 (Complete Rest) to 10 (Extremely Hard (almost maximal)). BORG CR10 was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
units on a scale
  Borg (Dyspnea) at Peak | 0.5 (0.4) | -0.3 (0.3)
  Borg (Dyspnea) at isotime | 0.4 (0.4) | -0.1 (0.3)
  Borg (Leg Effort) at Peak | -0.1 (0.3) | -0.3 (0.3)
  Borg (Leg Effort) at isotime: number analyzed (Participants) | 31 | 35
  Borg (Leg Effort) at isotime | 0.1 (0.3) | -0.2 (0.3)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; Borg (Dyspnea) at Peak: LSMeans, LSMean difference of CK-2127107 minus placebo, and 90% confidence intervals are based on a mixed effect model with treatment and period as fixed effects, subject as a random effect, and a compound symmetry covariance structure; Test type: Superiority; p = 0.099, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = -0.8, 90% CI 2-sided [-1.7 to 0.0]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; Borg (Dyspnea) at isotime: LSMeans, LSMean difference of CK-2127107 minus placebo, and 90% confidence intervals are based on a mixed effect model with treatment and period as fixed effects, subject as a random effect, and a compound symmetry covariance structure; Test type: Superiority; p = 0.255, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = -0.5, 90% CI 2-sided [-1.3 to 0.2]
Statistical Analysis 3: Comparison: Placebo vs CK-2127107; Borg (Leg Effort) at Peak: LSMeans, LSMean difference of CK-2127107 minus placebo, and 90% confidence intervals are based on a mixed effect model with treatment and period as fixed effects, subject as a random effect, and a compound symmetry covariance structure; Test type: Superiority; p = 0.651, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = -0.2, 90% CI 2-sided [-1.1 to 0.6]
Statistical Analysis 4: Comparison: Placebo vs CK-2127107; Borg (Leg Effort) at isotime: LSMeans, LSMean difference of CK-2127107 minus placebo, and 90% confidence intervals are based on a mixed effect model with treatment and period as fixed effects, subject as a random effect, and a compound symmetry covariance structure; Test type: Superiority; p = 0.591, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = -0.3, 90% CI 2-sided [-1.0 to 0.5]

7. Secondary Outcome: Change From Period Baseline at Week 2 in Respiratory Exchange Ratio (RER)
Description: The respiratory exchange ratio is equal to the VCO2 / VO2 [RER = VCO2 (L/min) / VO2 (L/min)]. RER was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
ratio
  Peak | -0.0036 (0.0125) | 0.0250 (0.0119)
  Isotime | -0.0042 (0.0102) | 0.0143 (0.0097)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.040, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.0286, 90% CI 2-sided [0.0061 to 0.0511]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.155, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean differencce = 0.0185, 90% CI 2-sided [-0.0031 to 0.0401]

8. Secondary Outcome: Change From Period Baseline at Week 2 in Carbon Dioxide Output (VCO2)
Description: VCO2 was defined as volume of CO2 exhaled from the body per unit of time; also called the rate of elimination of CO2. VCO2 was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
L/min
  Peak | -0.0129 (0.0231) | -0.0119 (0.0219)
  Isotime | -0.0115 (0.0188) | -0.0232 (0.0179)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.972, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.0010, 90% CI 2-sided [-0.0459 to 0.0479]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.578, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = -0.0118, 90% CI 2-sided [-0.0471 to 0.0236]

9. Secondary Outcome: Change From Period Baseline at Week 2 in End-tidal PCO2 (PETCO2)
Description: PETCO2 was defined as partial pressure of carbon dioxide in the expired gas at the end of an exhalation. This represents the mean partial pressure of carbon dioxide in the pulmonary alveoli. PETCO2 was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
mmHg
  Peak | -0.12 (0.34) | -0.77 (0.33)
  Isotime | -0.07 (0.33) | -0.64 (0.31)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.235, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = -0.65, 90% CI 2-sided [-1.55 to 0.26]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.215, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean differencce = -0.57, 90% CI 2-sided [-1.33 to 0.19]

10. Secondary Outcome: Change From Period Baseline at Week 2 in End-tidal PO2 (PETO2)
Description: PETO2 was defined as Partial pressure of oxygen in the expired gas at the end of an exhalation. This represents the mean partial pressure of oxygen in the pulmonary alveoli. PETO2 was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
mmHg
  Peak | 0.38 (042) | 1.08 (0.40)
  Isotime | 0.30 (0.40) | 0.75 (0.38)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.280, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.70, 90% CI 2-sided [-0.38 to 1.77]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.424, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.46, 90% CI 2-sided [-0.49 to 1.40]

11. Secondary Outcome: Change From Period Baseline at Week 2 in Tidal Volume (VT)
Description: VT was defined as tidal volume is the volume of gas exhaled in each respiratory cycle. Tidal volume is typically measured as an average value over several respiratory cycles, and is expressed in liters. VT was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
Liters
  Peak | -0.0689 (0.0216) | -0.0299 (0.0204)
  Isotime | -0.0582 (0.0289) | -0.0093 (0.0273)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.187, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.0390, 90% CI 2-sided [-0.0099 to 0.0879]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.213, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.0488, 90% CI 2-sided [-0.0163 to 0.1140]

12. Secondary Outcome: Change From Period Baseline at Week 2 in Breathing Frequency (Bf)
Description: Bf was defined as the number of breaths (i.e., an entire inspiratory and expiratory respiratory cycle) per minute. Bf was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Breaths/min
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 34
Breaths/min
  Peak | 1.6 (0.6) | 1.2 (0.6)
  Isotime | 1.4 (0.7) | 0.7 (0.7)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.640, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = -0.4, 90% CI [-2.1 to 1.2]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.487, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = -0.7, 90% CI 2-sided [-2.5 to 1.1]

13. Secondary Outcome: Change From Period Baseline at Week 2 in Inspiratory Capacity (IC)
Description: IC was defined as the volume of air that can be inspired after a normal expiration; it is the sum of the VT and the IRV. IC was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
Liters
  Peak | -0.047 (0.048) | 0.048 (0.046)
  Isotime | -0.09 (0.045) | 0.042 (0.043)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.100, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.095, 90% CI 2-sided [0.000 to 0.189]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.008, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.133, 90% CI 2-sided [0.053 to 0.213]

14. Secondary Outcome: Change From Period Baseline to Week 2 in Inspiratory Reserve Volume (IRV)
Description: The Inspiratory reserve volume was equal to VT - IC measured in liters [IRV (L) = VT (L) - IC (L)]. IRV was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
Liters
  Peak | 0.026 (0.049) | 0.077 (0.047)
  Isotime | -0.042 (0.050) | 0.052 (0.048)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.408, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.051, 90% CI 2-sided [-0.052 to 0.154]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.058, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.094, 90% CI 2-sided [0.013 to 0.174]

15. Secondary Outcome: Change From Period Baseline at Week 2 in Ventilatory Reserve (VE/MVV)
Description: VE/MVV provides the rate of expired ventilation to the capacity. VE/MVV was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: percentage of expired ventilation
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 34
percentage of expired ventilation
  Peak | 2.19 (2.18) | 3.62 (2.10)
  Isotime | 2.67 (2.34) | 3.52 (2.26)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.648, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 1.44, 90% CI 2-sided [-3.85 to 6.73]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.775, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.85, 90% CI 2-sided [-4.12 to 5.82]

16. Secondary Outcome: Change From Period Baseline at Week 2 in Heart Rate (HR)
Description: HR was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Beats/min
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
Beats/min
  Peak | -1.6 (1.5) | -0.5 (1.5)
  Isotime | -1.5 (1.7) | 0.7 (1.6)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.544, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 1.1, 90% CI 2-sided [-1.9 to 4.0]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.216, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 2.1, 90% CI 2-sided [-0.7 to 5.0]

17. Secondary Outcome: Change From Period Baseline at Week 2 in Systolic Blood Pressure (SBP)
Description: SBP was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data each specified time point.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
mmHg
  Peak | 3.0 (3.5) | -4.5 (3.3)
  Istotime | 0.2 (4.2) | 0.4 (4.0)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.171, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = -7.4, 90% CI 2-sided [-16.5 to 1.6]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.976, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.2, 90% CI 2-sided [-10.3 to 10.7]

18. Secondary Outcome: Change From Period Baseline at Week 2 in Diastolic Blood Pressure (DBP)
Description: DBP was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 32 | 35
mmHg
  Peak | 0.3 (2.1) | -0.3 (2.0)
  Isotime | -1.0 (2.0) | -2.0 (1.9)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.844, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = -0.6, 90% CI 2-sided [-6.1 to 4.9]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.751, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = -0.9, 90% CI 2-sided [-5.8 to 4.0]

19. Secondary Outcome: Change From Period Baseline at Week 2 in Arterial Oxygen Saturation From Pulse Oximetry (SpO2)
Description: SPO2 was defined as the noninvasive estimation of arterial hemoglobin (Hb) oxygen saturation, using a device that utilizes the combined principles of spectrophotometry and pulse plethysmography. SPO2 was reported at isotime and peak exercise during CWR test.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: percentage of oxygen saturation
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 31 | 34
percentage of oxygen saturation
  Peak | -0.4 (0.3) | -0.2 (0.2)
  Isotime | -0.3 (0.3) | 0.0 (0.2)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.590, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.2, 90% CI 2-sided [-0.5 to 0.9]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.399, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 0.3, 90% CI 2-sided [-0.3 to 0.9]

20. Secondary Outcome: Change From Period Baseline at Week 2 in Forced Vital Capacity (FVC)
Description: Change From Period Baseline in FVC was reported.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 33 | 34
Liters | 0.00 (0.05) | -0.10 (0.04)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.151, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = -0.09, 90% CI 2-sided [-0.20 to 0.01]

21. Secondary Outcome: Change From Period Baseline at Week 2 in Forced Expiratory Volume 1 (FEV1)
Description: Change From Period Baseline in FEV1 was reported.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 33 | 34
Liters | -0.030 (0.028) | -0.037 (0.027)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.857, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = -0.007, 90% CI 2-sided [-0.070 to 0.056]

22. Secondary Outcome: Change From Period Baseline at Week 2 in FVC/FEV1 Ratio
Description: Change From Period Baseline in FVC/FEV1 Ratio was reported.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 33 | 34
ratio | -1.10 (0.71) | 0.47 (0.69)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.110, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 1.56, 90% CI 2-sided [-0.05 to 3.17]

23. Secondary Outcome: Change From Period Baseline at Week 2 in Activation of Accessory Respiratory Muscles
Description: Activation of accessory respiratory muscles was assessed by electromyogram. Data was reported at peak and isotime.
Time Frame: Baseline and week 2 of each treatment period
Population: FAS population with available data at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: percentage of activation
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 31 | 32
percentage of activation
  Peak | 4.84 (4.76) | 6.91 (4.65)
  Isotime | 1.04 (4.39) | 3.98 (4.30)
Statistical Analysis 1: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.766, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 2.07, 90% CI 2-sided [-9.57 to 13.71]
Statistical Analysis 2: Comparison: Placebo vs CK-2127107; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.642, Mixed Models Analysis — Statistical comparison was performed at a 2-sided 0.10 significance level; LSMean difference = 2.94, 90% CI 2-sided [-7.66 to 13.54]

24. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: TEAEs were defined as any AE that started or worsened in severity after the first dose of study drug up to 14 days after the last dose of study drug. An AE was defined as any untoward medical occurrence in a participant administered a study drug or who had undergone study procedures and did not necessarily have a causal relationship with this treatment. An AE could therefore be any unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An abnormality identified during a medical test (e.g., laboratory parameter, vital sign, ECG data, physical examination) an AE only if the abnormality meets 1 of the following criteria: Induces clinical signs or symptoms, Requires active intervention, Requires interruption or discontinuation of study drug, The abnormality or test value is clinically significant in the opinion of the inves
Time Frame: From first dose of study drug up to 14 days after last dose of study drug (8 weeks)
Population: SAF population
Measure: Number; unit: Participants
Arm/Group | Placebo | CK-2127107
Number analyzed (Participants) | 41 | 42
Participants | 15 | 21

25. Secondary Outcome: Plasma Concentration of CK-2127107 at Day 1 Predose, Day 14 Lowest Concentration (Ctrough), and Day 14 Concentration Predose 6 Hours (C6h)
Description: Plasma concentration of CK-2127107 was reported.
Time Frame: Day 1 predose, day 14 Ctrough, day 14 C6h
Population: The pharmacokinetic analysis set (PKAS) consisted of the administered population for which ≥ 1 quantifiable plasma trough concentration or concentration at 6 hours was available for CK-2127107, or its metabolite CK-2127106.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | CK-2127107
Number analyzed (Participants) | 33
Nanogram per milliliter (ng/mL)
  Day 1 predose: number analyzed (Participants) | 17
  Day 1 predose | 0 (0)
  Day 14 Ctrough: number analyzed (Participants) | 32
  Day 14 Ctrough | 2620 (2100)
  Day 14 C6h | 3290 (2000)

26. Secondary Outcome: Plasma Concentration of CK-2127106 (Metabolite of CK-2127107) at Day 1 Predose, Day 14 Ctrough, Day 14 C6h
Description: Plasma concentration of CK-2127106 (metabolite of CK-2127107) was reported.
Time Frame: Day 1 predose, day 14 Ctrough, day 14 C6h
Population: PKAS population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CK-2127107
Number analyzed (Participants) | 33
ng/mL
  Day 1 predose: number analyzed (Participants) | 17
  Day 1 predose | 0 (0)
  Day 14 Ctrough: number analyzed (Participants) | 32
  Day 14 Ctrough | 1760 (1710)
  Day 14 C6h | 1770 (1620)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 14 days after last dose of study drug (8 weeks)
Arm/Group | Placebo | CK-2127107
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/41 | 2/42
Other Adverse Events (participants affected / at risk) | 1/41 | 3/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=41) | CK-2127107 (N=42)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=41) | CK-2127107 (N=42)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT02662582/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT02662582/SAP_001.pdf